CLINICAL TRIAL: NCT04530682
Title: Seroprevalence and Clinical Expression of SARS-CoV-2 Infection in Patients With Chronic Inflammatory Rheumatisms and Impact of Immuno-suppressive Drugs on the Persistence of Anti-SARS-CoV2 Antibodies During Two Years of Follow-up
Brief Title: COVID-19 in Rheumatic Inflammatory Diseases Under Immuno-suppressive Drugs
Acronym: COVIDRIC-2
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: French Society of Rheumatology (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0409; UF8074 (Other: Montpellier University Hospital)
Record Dates: First submitted 2020-07-27; First posted 2020-08-28 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Chronic Inflammatory Rheumatism
Keywords: COVID-19; SARS-CoV2; Rheumatoid arthritis; Spondyloarthritis; Seroprevalence; Seropersistence
MeSH Terms: conditions — COVID-19; Arthritis, Rheumatoid; Spondylarthritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and plasma samples at baseline. Serum samples at 0, 6, 12 and 24 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SARS-CoV-2 seropositive patients with chronic inflammatory rheumatisms (CIRs): 200 SARS-CoV-2 seropositive patients with chronic inflammatory rheumatisms (CIRs) from the COVID-RIC-1 cohort.
  Interventions: Biological: Biological samples
- Control group: 100 health professionals participating in the COVID-BIOTOUL cohort will be selected to be matched on age, gender, and the time between the date of infection with Covid-19 and the first serology of CIR patients.

INTERVENTIONS:
Biological: Biological samples — Serum and plasma samples. At baseline, 6, 12 and 24 months
  Groups: SARS-CoV-2 seropositive patients with chronic inflammatory rheumatisms (CIRs)

SUMMARY:
Accurate knowledge of the humoral immune responses induced by SARS-CoV-2 in patients undergoing immunosuppressive therapy is essential to guide recommendations for infected patients and for vaccination policy for uninfected immunosuppressed patients.

DETAILED DESCRIPTION:
Longitudinal, cas-control study, observational multicenter study based on a cohort of 200 SARS-CoV-2 seropositive patients with chronic inflammatory rheumatisms (CIRs) from the COVID-RIC-1 cohort.

The follow-up the persistence of SARS-CoV-2 serological status for 2 years in 200 patients with inflammatory rheumatisms compared to matched 100 healthy controls to evaluate the impact of immuno-suppressive therapy will be proposed.

Schedule: 4 visits over a 24-month period.

An observational routine care study was initiated in 16 French hospitals to assess the SARS-CoV-2 seroprevalence in France in a population with CIRs (Covid-RIC-1). The project plans to screen 5000 CIRs patients. The COVID-RIC-2 study will thus be proposed to these pre-screened subjects according to their positive status in the serology for SARS-CoV-2 at the time of their inclusion in COVID-RIC-1.

For the control group, 100 health professionals participating in the COVID-BIOTOUL cohort will be selected to be matched on age, gender, and the time between the date of infection with Covid-19 and the first serology of CIR patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with rheumatoid arthritis or spondyloarthritis
* With positive serology for SARS-CoV-2 infection less than 3 months old at the time of inclusion
* Under biotherapy, or conventional synthetic Disease-modifying antirheumatic drugs (csDMARD) or Nonsteroidal anti-inflammatory drugs (NSAIDs) or steroids for at least one month during the year 2020
* Agreeement to participate two years in the study

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 200 participants with chronic inflammatory rheumatisms and positive status in the serology for SARS-CoV-2. This population will be compared with a healthy control group from the cohort Covid-Biotoul
Sampling Method: Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2022-06-23 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Distribution of anti-SARS-CoV-2 neutralising immunoglobulin titres in patients with chronic inflammatory rheumatisms | at baseline
  Distribution of anti-SARS-CoV-2 neutralising immunoglobulin titres at baseline in patients with chronic inflammatory rheumatisms
Distribution of anti-SARS-CoV-2 neutralising immunoglobulin titres in patients with chronic inflammatory rheumatisms | at 6 months after inclusion
  Distribution of anti-SARS-CoV-2 neutralising immunoglobulin titres at 6 months in patients with chronic inflammatory rheumatisms

SECONDARY OUTCOMES:
To assess the maintenance of SARS-CoV-2 seroconversion in patients with chronic inflammatory rheumatisms (CIRs) compared to non-CIR controls. | at 12 months after inclusion
  To assess the maintenance of SARS-CoV-2 seroconversion at 12 months in patients with CIRs compared to non-CIR controls.
To assess the maintenance of SARS-CoV-2 seroconversion at 24 month in patients with chronic inflammatory rheumatisms (CIRs) compared to non-CIR controls | at 24 months after inclusion
  To assess the maintenance of SARS-CoV-2 seroconversion at 24 months in patients with CIRs compared to non-CIR controls.
Assess the impact of the pandemic and its consequences on the psychological state of patients with chronic inflammatory rheumatisms | baseline
  Assess the impact at baseline of the pandemic and its consequences on the psychological state of patients with chronic inflammatory rheumatisms using different validated questionnaires
Assess the impact of the pandemic and its consequences on the psychological state of patients with chronic inflammatory rheumatisms | at 6 month after inclusion
  Assess the impact at 6 month of the pandemic and its consequences on the psychological state of patients with chronic inflammatory rheumatisms using different validated questionnaires
Assess the impact of the pandemic and its consequences on the psychological state of patients with chronic inflammatory rheumatisms | at 12 month after inclusion
  Assess the impact at 12 month of the pandemic and its consequences on the psychological state of patients with chronic inflammatory rheumatisms using different validated questionnaires
Assess the impact of the pandemic and its consequences on the psychological state of patients with chronic inflammatory rheumatisms | at 24 month after inclusion
  Assess the impact at 24 month of the pandemic and its consequences on the psychological state of patients with chronic inflammatory rheumatisms using different validated questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- Centre hopsitalier universitaire de Montpellier, Montpellier, Occitanie, France